CLINICAL TRIAL: NCT05845970
Title: An Investigation Into the Efficacy of a Botanical Supplement to Provide Period Relief
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Focus Consumer Healthcare (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20268
Record Dates: First submitted 2023-04-03; First posted 2023-05-06 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Menstrual Pain; Premenstrual Syndrome
MeSH Terms: conditions — Dysmenorrhea; Premenstrual Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Single Group (Experimental): Single-group crossover trial with 100 total participants. Participants will use Pamprin Botanicals during their first period and both Pamprin Botanicals and over-the-counter Pamprin Menstrual Relief during their second period.
  Interventions: Other: Pamprin Botanicals; Combination Product: Pamprin Botanicals + Pamprin Menstrual Pain Relief

INTERVENTIONS:
Other: Pamprin Botanicals — Participants will take Pamprin Botanicals only. Participants will take 450mg of Pamprin Botanicals two days before their predicted period and then take it every day during their period. Participants can also take Pamprin Botanicals two days after the bleeding has concluded.
Combination Product: Pamprin Botanicals + Pamprin Menstrual Pain Relief — Participants will repeat taking Pamprin Botanicals two days before their second predicted period and continue to take it each day during their period. However, during the second period, participants will also take Pamprin Menstrual Pain Relief per the over-the-counter directions (2 tablets every 6 hours with water).

SUMMARY:
Women often experience significant pain during their periods which can significantly impact on quality of life. In this study, two products that are used to alleviate period pain will be examined. One test product is botanically based, and the other is a traditional over-the-counter pain reliever with additional components added to support less painful periods. The trial will be a cross-over trial where participants will use the botanical product before, during, and after their first period. Participants will use the botanical product alongside a traditional over-the-counter period product during their second period. Participants will answer surveys and have blood drawn at a third-party lab to answer the main objectives of this trial.

ELIGIBILITY:
Inclusion Criteria:

* Female between 18-40 years of age.
* Must be in good health with no significant chronic conditions and a BMI under 35.
* Must experience period pain and other PMS symptoms.
* Must have a regular menstrual cycle with a bleed week.
* If using hormonal contraception, must do so for at least three months
* If using oral contraception, must allow for bleed week.
* Must be able to predict their bleed week.
* Willing to abstain from strenuous exercise 24 hours before each of the three blood draws in this trial.

Exclusion Criteria:

* Suffers from pre-existing conditions that would prevent them from adhering to the protocol.
* Anyone with known severe allergic reactions.
* Anyone with a previous negative experience with acetaminophen.
* Unwilling to follow the study protocol.
* Currently pregnant, breastfeeding, or wanting to become pregnant for the duration of the study.
* Anyone who uses other supplements for period pain and PMS symptoms.
* Current use of an extended activity hormonal contraception (examples include Depo-provera or Nexplanon.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2023-02-08 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Changes in common menstrual cycle symptoms [Time Frame: 2 menstrual cycles (approximately 60 days)] | 60 days
  Menstrual cycle symptoms will be measured via study-specific questionnaires.

SECONDARY OUTCOMES:
Changes in blood biomarkers during the menstrual cycle [Time Frame: 2 menstrual cycles (approximately 60 days)] | 60 days
  hs-CRP and cortisol will be measured via blood draws. Blood draws will occur at Baseline, Day 5 of bleeding during their first menstrual cycle during the study, and Day 5 of bleeding during their second menstrual cycle during the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Santa Monica, California, United States